CLINICAL TRIAL: NCT04817605
Title: Effects of Therapeutic Exercise in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Sandra Jiménez, University of Valladolid Faculty of Health Sciences, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVa
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Therapeutic Exercise; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Therapy (Experimental)
  Interventions: Other: Therapeutic Exercise

INTERVENTIONS:
Other: Therapeutic Exercise — Exercise therapy based primarily in aerobic exercise according clinical guidelines last recommendations.To perform different whole body aerobic exercises with a mild to moderate intensity according to Borg scale and maximum heart rate.

SUMMARY:
Fibromyalgia syndrome is characterized by chronic generalized musculoskeletal pain associated with fatigue, sleep disturbances and some biochemical markers. The European League Againts Rheumatism (EULAR) described an algorithm how to treat step by step these patients.

The objective of this trial is to evaluate if therapeutic exercise is effective on fatigue, pain threshold, quality of life, quality of sleep, pain coping and biochemical and genetic markers.

For this purpose, the investigators conduct a randomized controlled trial double-blind (patient and examiner). The investigators included patients diagnosed of fibromyalgia according to the American College of Rheumatology (ACR).

Patients included one group receiving exercise therapy consisting of 3 treatment sessions a week over 10 weeks.

The variables are measured at the beginning and end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed medically with Fibromyalgia
* Diagnosed according to the American College of Rheumatology criteria
* Agreement to attend to treatment sessions

Exclusion Criteria:

* Any kind of contraindications for physical activity
* Other kind of diseases that could limit the intervention
* Previous surgery last year
* Medication modifications in the last 3 months

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Baseline
  VAS
Pain intensity | through study completion, an average 10 weeks
  VAS
Quality of Sleep | Baseline
  The investigators measure the quality of sleep with Pittsburg Sleeping Questionnaire Index (PSQI) at baseline
Quality of Sleep | through study completion, an average 10 weeks
  The investigators measure the quality of sleep with Pittsburg Sleeping Questionnaire Index (PSQI) at baseline

SECONDARY OUTCOMES:
Pressure pain threshold | Baseline
  The investigators measure the pressure pain threshold of the 18 points described initially by the American College of rheumatology with a digital algometer at baseline
Pressure pain threshold | through study completion, an average 10 weeks
  The investigators measure the pressure pain threshold of the 18 points described initially by the American College of rheumatology with a digital algometer at the end of treatment
Central sensitization | Baseline
  The investigators measure the central sensitization with Chronic Pain Self-Efficacy Scale (CPSS) at baseline
Central sensitization | through study completion, an average 10 weeks
  The investigators measure the central sensitization with Chronic Pain Self-Efficacy Scale (CPSS)
Analysis of tryptophan metabolites | Baseline
  The investigators measure the tryptophan metabolites with blood test analysis at baseline
Analysis of tryptophan metabolites | through study completion, an average 10 weeks
  The investigators measure the tryptophan metabolites with blood test analysis at baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Sandra Jiménez Jiménez-del-Barrio, Soria, Spain

IPD SHARING:
Plan to Share IPD: Undecided